CLINICAL TRIAL: NCT02428413
Title: Evaluation and Control of Waste Anesthetic Gas (WAG) in the Post Anesthesia Care Unit (PACU) Within Patient and Caregiver Breathing Zone
Brief Title: Evaluation and Control of WAG in PACU Within Patient and Caregiver Breathing Zone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Teleflex (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2015-05
Record Dates: First submitted 2015-04-16; First posted 2015-04-28 (Estimated); Results first posted 2016-09-29 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-08

CONDITIONS: Waste Anesthetic Gas (WAG) Emanating From Patients Post-operative Recovery
Keywords: Waste Anesthetic Gas (WAG)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard oxygen mask (Active Comparator): Standard face mask to provide supplemental oxygen
  Interventions: Device: Standard oxygen mask
- ISO-Gard Mask (Active Comparator): Face mask to scavenge waste anesthetic gases from patient during recovery from general anesthesia and to provide supplemental oxygen.
  Interventions: Device: ISO-Gard Mask

INTERVENTIONS:
Device: ISO-Gard Mask — to scavenge waste anesthetic gases from patients and provide supplemental oxygen
  Arms: ISO-Gard Mask
Device: Standard oxygen mask — Provide supplemental oxygen
  Arms: Standard oxygen mask

SUMMARY:
The purpose of this study is to evaluate anesthetic gas in the PACU within patient and caregiver breathing zones.

DETAILED DESCRIPTION:
The purpose of this single-center, multi-arm, randomized controlled study is to evaluate use of the ISO-Gard mask in patients immediately following a surgical procedure in which inhaled anesthetic is used as the primary modality of anesthesia, for the following: 1) measure the waste anesthetic gas emanating from patient during the immediate one hour post-operative recovery period in the PACU; 2) measure waste anesthetic gas within PACU caregiver's breathing zone; and 3) determine the efficacy of the ISO-Gard mask in reducing caregiver's exposure to waste anesthetic gas in the PACU.

Subjects who will receive either Sevoflurane or Desflurane inhaled anesthetic will be enrolled in this study. Subjects will be randomized to receive either the ISO-Gard scavenging mask or a traditional supplemental oxygen mask post operatively; all other elements of the subjects' care will be in accordance with the institution's standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18-120 years of age.
* Patients requiring inhaled anesthetic agents as part of their anesthesia during surgery (Sevoflurane or Desflurane)
* Patients with following outpatient procedures scheduled for a duration of greater than 2 hours per the operating room schedule:

  1. . Bariatric procedures
  2. Robotic surgery cases
  3. Orthopedic
  4. Gynecological procedures
  5. ENT
  6. Plastic
* Not documented as terminally ill
* Subject expected to remain in PACU for at least one hour
* Subject or legally authorized representative has provided written informed consent prior to the procedure using a form that is approved by the Institutional Review Board (IRB).

Exclusion Criteria:

* Patients are/were given/planned to be given total IV anesthetics during surgery
* Any patient that is not expected to tolerate a mask in PACU
* Subject has already been enrolled in study
* Subject is an employee of the Investigator or has involvement in other studies under the direction of investigator or study site
* Women who are pregnant
* End of anesthetic gas administration in PACU bay greater than 45 minutes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2015-04; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W Williams III, MD, Principal Investigator — U of Texas Medical school at Houston

IPD SHARING:
Plan to Share IPD: Yes
The aggregate study results will be reported collectively, not individually by participant.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patient screening took place in the day surgery unit at Memorial Hermann Hospital in the Texas Medical Center of Houston Texas between July 2015 and November 2015.
Period: Overall Study
Arm/Group | Standard Oxygen Mask | ISO-Gard Mask
Started | 64 | 61
Completed | 56 | 52
Not Completed | 8 | 9
Not completed — Device to measure WAG malfunctioned | 3 | 5
Not completed — Protocol Violation | 1 | 2
Not completed — Case Cancelled | 2 | 0
Not completed — Missed Cases | 1 | 2
Not completed — Nurse Refusal | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Oxygen Mask | ISO-Gard Mask | Total
Number analyzed (Participants) | 56 | 52 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 49 | 42 | 91
  >=65 years | 7 | 10 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 28 | 69
  Male | 15 | 24 | 39

OUTCOME MEASURES:

1. Primary Outcome: Waste Anesthetic Gas Measured by Parts Per Million Within PACU Caregiver's Breathing Zone With Caring for Patients
Description: The measurement of Waste Anesthetic Gas in parts per million resolution emanating from the patient to the caregiver's breathing zone.
Time Frame: 1 hour post-operative recovery period
Population: A study size of 100 randomized subjects will be used. Aforementioned sample size was determined to be able to detect an effect size of 0.57 that would provide 80% power and 5% type I error (95% confidence interval and p-0.05 level of significance). Two sample student t-test will be used to do data analysis.
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Standard Oxygen Mask | ISO-Gard Mask
Number analyzed (Participants) | 56 | 52
parts per million | 60.6 (20.6) | 56.9 (9.7)
Statistical Analysis 1: Comparison: Standard Oxygen Mask vs ISO-Gard Mask; Test type: Superiority or Other; p = 0.24, t-test, 2 sided

2. Primary Outcome: Waste Anesthetic Gas Measured by Parts Per Million Emanating From Patients During Normal PACU Working Conditions
Description: The measurement of Waste Anesthetic Gas in parts per million emanating from the patient between the standard oxygen mask and the ISO-Gard oxygen mask.
Time Frame: 1 hour post-operative recovery period
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Standard Oxygen Mask | ISO-Gard Mask
Number analyzed (Participants) | 56 | 52
parts per million | 58.7 (8.1) | 56.7 (10.2)
Statistical Analysis 1: Comparison: Standard Oxygen Mask vs ISO-Gard Mask; Test type: Superiority or Other; p = 0.26, t-test, 2 sided

3. Primary Outcome: Efficacy of the ISO-Gard Mask in Reducing Caregiver's Exposure to WAG-Percentage of Time
Description: For MAX-WAG measurements obtained every 30 seconds, we calculated the percentage of time in MAX-WAG [>2ppm] relative to the total collection period.
Time Frame: 1 hour post-operative recovery period
Measure: Median (Inter-Quartile Range); unit: percentage of time
Arm/Group | Standard Oxygen Mask | ISO-Gard Mask
Number analyzed (Participants) | 56 | 52
percentage of time | 5.2 [2.4 to 10.4] | 2.0 [0 to 5.7]

4. Primary Outcome: Efficacy of the ISO-Gard Mask in Reducing Caregiver's Exposure to WAG-Duration
Description: For MAX-WAG measurements obtained every 30 seconds, we calculated the duration of MAX-WAG [>2ppm]
Time Frame: 1 hour post-operative recovery period
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | Standard Oxygen Mask | ISO-Gard Mask
Number analyzed (Participants) | 56 | 52
minutes | 3.0 [1.5 to 6.5] | 1.0 [0 to 3.0]

ADVERSE EVENTS:
Arm/Group | Standard Oxygen Mask | ISO-Gard Mask
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/52
Other Adverse Events (participants affected / at risk) | 0/56 | 0/52

LIMITATIONS AND CAVEATS:
Precise dosing of anesthetic gas was not recorded. Dosing is practitioner dependent. Duration of surgery, PACU nurse interactions with patients, including proximity, attention to patient, and number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less